CLINICAL TRIAL: NCT02490241
Title: Lithium Therapy: Understanding Mothers, Metabolism and Mood
Acronym: LiThiUM
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Crystal Clark, Associate Professor, Northwestern University
Other Study IDs: 00200026
Record Dates: First submitted 2015-05-26; First posted 2015-07-03 (Estimated); Last update posted 2022-10-05 (Actual); Status verified 2022-10

CONDITIONS: Bipolar Disorder
Keywords: pregnant; female; women; lithium; bipolar
MeSH Terms: conditions — Bipolar Disorder | interventions — Lithium; Lithium Carbonate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood serum specimen will be obtained to measure lithium levels. Urine will be collected to measure lithium levels and creatinine clearance. Standard of care labs will be obtained on every participant that is eligible and signs informed consent. Participants will also have the option to have blood drawn for DNA banking.
  Participants in the study that elect to receive analgesia for pain related to labor and have a spinal-epidural at Northwestern University will have CSF stored and banked for future analysis.
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Lithium — Patients taking lithium as a mood stabilizer during pregnancy are eligible to participate in the study. Their dose and serum concentration levels of lithium will be monitored throughout pregnancy and up to three months postpartum.
  Other Names: lithium carbonate

SUMMARY:
Lithium, the gold standard for treatment of Bipolar Disorder (BD) and a common augmentation to medication therapy for Major Depression, is commonly continued in pregnancy due to its therapeutic benefit and more recent data that suggests the teratogenic effects of lithium are less than historically believed. Due to the increased elimination of lithium during pregnancy, lithium concentration decreases in the blood and women with BD are vulnerable to BD episode recurrence in pregnancy. Uncontrolled symptoms of BD in pregnancy increase the risk for postpartum exacerbation of BD and psychosis. Our study will investigate the pharmacokinetics (PK) of lithium prior to pregnancy, during pregnancy, and postpartum. Twenty women taking lithium in pregnancy or planning to become pregnant and continue lithium will be invited to participate in a study to measure repeated blood levels of lithium at six time points between preconception and 3 months postpartum. The data collected will inform the dose, timing of dose, and frequency of dosing of lithium that will lead to fewer untoward effects for the mother and baby. Change in elimination clearance of lithium will be correlated with symptom worsening to develop a dosing algorithm that will help maintain wellness for pregnant women with mood disorders.

DETAILED DESCRIPTION:
There is an increased risk of recurrence of Bipolar Disorder (BD) episodes or worsening symptoms in pregnancy after the discontinuation of mood stabilizers. Similarly, changes in medication concentration due to the physiological changes in pregnancy may effectively reduce the medication dose and thus its efficacy in pregnancy. Therapeutic dose monitoring has proven to have great utility in preventing seizure recurrence in women with epilepsy (WWE). Similar guidelines to that of women with epilepsy would benefit pregnant women with BD who are taking mood stabilizing medications in pregnancy. Current evidence suggests that lithium has a more favorable reproductive profile than many mood stabilizing antiepileptic agents. However, the pharmacokinetics as well as the utility of therapeutic dose monitoring of lithium in pregnant patients with Bipolar Disorder has not been well studied.

This study is an observational protocol to explore the longitudinal pharmacokinetics (PK) of lithium during pregnancy and postpartum in 20 women with Bipolar Disorder. The correlation between changes in bioavailability and concentrations ratios and increases in symptoms of depression, mania and anxiety and recurrence of syndromal BD episodes that fulfill Diagnostic and Statistics Manual of Mental Disorders (IV) (DSM4) criteria will be investigated.

The primary aims of this study are 1.) To describe the changes in lithium elimination and serum concentration across pregnancy and postpartum to establish its efficacious use and dosing requirements during childbearing 2.) To evaluate the associations between maternal and umbilical cord lithium serum levels. 3.) To explore the relationship between declining lithium serum concentrations during pregnancy and the increase in psychiatric symptoms and recurrence of syndromal BD.

To optimize the research yield from this investigation, participants will have the option to allow banking of cerebrospinal (CSF) fluid and DNA for future analyses.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* If Pregnant, equal to or less than 26 weeks
* English-speaking
* DSM-IV Bipolar Disorder, any subtype, Major Depressive Disorder, or Mood Disorder Not Otherwise Specified
* Able to provide informed consent
* Daily dosing of lithium

Exclusion Criteria:

* Active substance abuse within last 6 months and/or positive urine drug screen
* Active suicidality
* No obstetrical care
* Use of other drugs that affect metabolism of lithium
* Medications in FDA categories F or X that are not antimanic drugs
* Chronic Kidney Disease

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pre-conception planning and pregnant women taking lithium for the purpose of mood stabilizing will be recruited broadly from Northwestern clinical services, including Internal Medicine, OB/GYN, Family Medicine, and Psychiatry, registries, and from the local Chicagoland community. Patients that sign consent, complete the evaluation and meet criteria will be enrolled into the study.
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2015-04; Primary Completion 2019-12 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
Change in Serum concentration/elimination | An average of every 10 weeks, beginning at the preconception visit where a baseline concentration level will be established, at 3 timepoints throughout pregnancy, and at two and twelve weeks postpartum
  For patients on 1x day dosing, serum levels will be obtained beginning at time 0 and at hours, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, and 24 and L/D ratio will be determined at each time point. This series of serum levels will be completed an average of every 10 weeks across pregnancy, and postpartum. For patients on 2x dosing, serum levels will be obtained at time 0 and at hours 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, and 12.
  All urine excreted during participant's overnight research visits will be collected to perform lithium and creatinine clearance tests.

SECONDARY OUTCOMES:
Infant (umbilical cord)/Maternal ratio of lithium | 30 min
  Ratio of umbilical cord (infant) lithium serum level to maternal lithium serum level will be determined at delivery.
Scores on Depression assessment, Inventory of Depression Symptomatology- Self Report (IDS-SR) | Participants will complete these assessments an average of every 10 weeks from the time they enter the study, up to 12 weeks postpartum
  To determine if there is a pattern of increasing scores on self-report depression assessment (IDS-SR) and declining L/D ratios. Increasing scores indicate worsening symptoms or depression episode recurrence.
Scores on mania assessment, Young Mania Reporting Scale (YMRS) | Participants will complete these assessments an average of every 10 weeks from the time they enter the study, up to 12 weeks postpartum.
  To determine if there is a pattern of increasing scores on clinician administered mania assessment (YMRS) and declining L/D ratios.
Scores on anxiety scale, Generalized Anxiety Disorder (GAD-7) | Participants will complete these assessments an average of every 10 weeks from the time they enter the study, up to 12 weeks postpartum.

CONTACTS AND LOCATIONS:
Overall Officials: Crystal T Clark, MD, MSc, Principal Investigator — Northwestern University
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No